CLINICAL TRIAL: NCT00845013
Title: Epidemiology and Pathogenesis of HIV-Associated Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: HIVPAP
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: HIV Infection; Pulmonary Hypertension; Endothelial Function; HIV Infections
Keywords: HIV infection; pulmonary hypertension; endothelial function; antiretroviral medication; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, PBMCS, BAL
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV Infection: HIV-infected individuals with the clinical diagnosis of pulmonary hypertension or HIV-infected individuals who have mildly elevated pulmonary arterial pressures

SUMMARY:
The purpose of this study is to describe the epidemiology of pulmonary hypertension in individuals with HIV infection and to investigate its pathogenesis. We propose to conduct a prospective observational cohort study to determine the association between highly active antiretroviral therapy (HAART) and viral suppression in HIV-infected patients who have been identified to have pre-clinical pulmonary hypertension (Aim 1). In addition, we will investigate the mechanistic role of the HIV-1 Nef protein and HHV-8 infection in the development and progression of pulmonary hypertension in individuals with HIV (Aim 2). We will also investigate endothelial function in HIV-infected patients with pulmonary hypertension (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

1. Infection with HIV greater than 6 months in duration
2. Right heart catheterization showing PASP > 30mm Hg
3. Ability to provide reliable history of HIV medications or has received the majority of medical care from San Francisco General Hospital with available records of medical treatment.
4. Ability to participate in follow-up for the duration of the study.

Exclusion Criteria:

1. Known significant cardiovascular disease, including clinically significant valvular heart disease, congenital heart disease, current or prior symptomatic coronary disease, or known cardiomyopathy.
2. Any known pulmonary disease that could potentially cause pulmonary hypertension.
3. A pO2 by pulse oximetry below 90% on room air.
4. Obstructive sleep apnea.
5. Known collagen vascular disease.
6. History of anorexigen use

   * 7. Age less than 18 years old.
   * 8. Other co-morbidities for which the investigators, in conjunction with the primary care provider, believe render the participant with an expected survival of 6 months or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected individiuals with the clinical diagnosis of pulmonary hypertension or who have mildly elevated pulmonary arterial pressures
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2007-11; Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
pulmonary artery pressure | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No